CLINICAL TRIAL: NCT07203014
Title: Testing a Brief, Engagement Focused Intervention for Parents and Educators in Preschool: Parent-Educator Action Response
Brief Title: Parent-Educator Action Response
Acronym: PEAR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Courtney Zulauf-McCurdy, Assistant Professor, Pritzker Department of Psychiatry and Behavioral Health, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000176; K23MH129575 (NIH)
Record Dates: First submitted 2025-09-22; First posted 2025-10-02 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders
Keywords: adjunctive intervention; Preschool ADHD symptoms; Disruptive Behavior; Parent-teacher relationship; Daily Report Card
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Problem Behavior

STUDY DESIGN:
Intervention Model Description: The study uses a pilot roll-out implementation optimization (ROIO) design. A ROIO is a novel methodological innovation that provides a rigorous solution to optimization via iterative, rapid incorporation of partner input throughout implementation in pursuit of effective, affordable, scalable, and efficient outcomes.
  There will be three clusters over the course of the trial. Each cluster will contain 1-3 early childhood centers. Teachers from each classroom within each center will be recruited and 1-4 families will be recruited from each classroom that has a participating teacher. All participants will receive information on the Daily Report Card followed by the new adjunctive intervention (PEAR). There is no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEAR intervention group (Experimental): All participants will receive the Daily Report Card plus PEAR. PEAR is delivered via group sessions in which participants will be guided through content with a licensed clinical psychologist and will complete activities and receive handouts for reference.
  Interventions: Behavioral: Parent-Educator Action Response (PEAR); Behavioral: Daily Report Card

INTERVENTIONS:
Behavioral: Parent-Educator Action Response (PEAR) — PEAR is a novel adjunctive intervention aimed at improving teacher and family implementation of classroom-based interventions for child ADHD symptoms and disruptive behavior in preschool.
Behavioral: Daily Report Card — The Daily Report Card is a behavioral intervention for children with challenging behaviors, and provides a structure for teachers and caregivers to support a child with reducing challenging behaviors and increasing positive behaviors. The DRC has been shown to be highly effective in reducing ADHD symptoms.

SUMMARY:
The goal of this clinical trial is to learn if a new adjunctive intervention, Parent-Educator Action Response (PEAR), works to improve teacher and family engagement in school-based interventions for child attention deficit/hyperactivity disorder (ADHD) and disruptive behavior symptoms. This clinical trial will also be used to refine implementation procedures to inform a larger clinical trial.

DETAILED DESCRIPTION:
School-based behavioral interventions are well-established treatments for preschool children who display elevated ADHD symptoms, regardless of a diagnosis, and are the recommended first line of treatment according to the American Academy of Pediatrics. However, teachers and families face barriers to implementing behavioral interventions with the recommended frequency and fidelity. The investigators are proposing to test a new adjunctive intervention that is aimed at improving teacher and family implementation of school-based interventions for preschool disruptive behavior and ADHD symptoms. The investigators will be testing PEAR plus a school-based intervention (Daily Report Card; DRC) in a pilot roll-out implementation optimization (ROIO) trial with three clusters (groups of schools) across two years.

Adjunctive Intervention (PEAR). All participating parents and teachers will complete PEAR. PEAR consists of three group sessions (one for caregivers and one for educators) followed by a meeting with each caregiver-educator dyad.

Daily Report Card. The primary goal of PEAR is to improve teacher and family implementation of an evidence-based practice for ADHD symptoms in preschool. The investigators have decided to focus on implementation of the Daily Report Card. Following consent, teachers will receive handouts on the Daily Report Card and will be asked to implement it for the child whose parents are in PEAR. Teachers and parents will be asked to complete weekly reports measuring teacher and family daily use of the DRC starting at BL through the 4-week follow up (8 weeks total).

Assessment Procedures. Assessments will be completed at three time points: BL (week 0), post-PEAR (4 weeks from BL), and follow-up (8 weeks from BL). At each assessment, participating legal guardians and teachers will complete rating scales electronically via RedCap, a scalable, secure, enterprise-level application for data collection. Interviews: Qualitative interviews with parents and teachers who participate in PEAR will be conducted to understand their experiences and identify potential areas for improvement.

Analytic Approach. This clinical trial will specifically examine the acceptability, feasibility and promise of PEAR and refine and optimize trial procedures. Basic data screening and descriptive analyses will be conducted for all variables, and the investigators will screen for errors, distributional form, and missing data. For all models, the investigators will check assumptions to ensure that results are not an artifact of violations. Below are analytic details for each aim of the trial:

Is PEAR and the implementation strategies acceptable and feasible? Overall, PEAR acceptability and feasibility for all participants will be evaluated by examining the mean parent and teacher ratings of satisfaction, acceptability, appropriateness, and feasibility. Consumer fit will be considered acceptable if scores are above the neutral point of the scale for all measures except fidelity, which the investigators will consider 80% as the target point. The investigators will also examine whether acceptability and feasibility indices vary by classroom and participant demographics by treating these predictors as fixed effects in regression analyses.

Are the ROIO trial procedures acceptable and feasible? This aim is focused on (a) refining recruitment procedures and study protocol to obtain an adequate sample of parents, (b) optimizing screening and assessment procedures in preschool, and (c) optimizing procedures for sustaining participants in PEAR (i.e., minimizing drop-out).

Does PEAR improve teacher and family fidelity to the Daily Report Card? The investigators will collect daily (weekdays only) counts of family and teacher implementation of the Daily Report Card starting at BL through follow-up (8 weeks total). Fidelity will be defined as the proportion of weekdays the Daily Report Card is implemented at home, school, and both. The investigators are interested in examining the change in fidelity across time. Hierarchical multi-level models will be used to ensure inclusion of random effects, variations between clusters, variation between times within cluster, and fixed effects of time which will be estimated independently of treatment effect, so that systematic change over time will not be mistaken for the effect of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Teacher or legal guardian/caregiver of a preschool-aged child between 2-5 years old
* Child has behavioral challenges in the classroom or needs support with social-emotional development
* Teacher participants must be fluent in English
* Caregiver participants may be fluent in English or Spanish.

Exclusion Criteria:

* Teacher or legal guardian/caregiver of a child who is not 2-5 years old
* Child does not have behavioral challenges or does not need support with social-emotional development
* Teacher participants who are not fluent in English
* Caregiver participants who are not fluent in either English or Spanish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Daily Report Card Check-In | Baseline to 8-week follow-up
  The Daily Report Card (DRC) check-in is a weekly survey developed by the investigators that measures daily uptake of DRC usage among parents and teachers across home and school.

SECONDARY OUTCOMES:
Preschool Pediatric Symptom Checklist | Baseline, 4-week, 8-week follow-ups.
  Teachers and parents will complete the Preschool Pediatric Symptom Checklist (Sheldrick et al., 2012) to evaluate overall child behavior. The Preschool Pediatric Symptom Checklist is an 18-item scale with answer choices of 0 = Not at all to 2 = Very much. Items are summed to obtain a score; authors recommend a clinical cutoff score of 9 (highest possible score is 36).
Preschool ADHD Rating Scale Version IV (ADHD-RS-IV) | Baseline, 4-week, 8-week follow-ups.
  Teachers and parents will complete the Preschool ADHD-RS-IV to measure child ADHD symptoms of children 3-5 years old. The Preschool ADHD-RS-IV (McGoey et al., 2007) is an 18-item scale with answer choices from 0 = rarely or never to 3 = very often. Total score is the sum of all 18 items, odd numbered items measure inattention and even numbered items measure hyperactivity/inactivity. 93rd percentile cutoff scores for boys are as follows: 32 (parent) and 38 (teacher); 93rd percentile cutoff scores for girls are as follows: 24 (parent) and 24 (teacher).
Teacher-Parent Alliance | Baseline, 4-week, 8-week follow-ups.
  Teachers and parents will complete an adapted version of the Working Alliance Inventory - Short Revised (WAI-SR; Hatcher & Gillaspy, 2006) to measure teacher-parent alliance. The investigators adapted this measure to better fit the context. The 12-item measure uses a 5-point Likert scale from 1 = seldom to 5 = always.
Teacher-Parent Joining | Baseline, 4-week, 8-weeks follow-ups.
  Teachers and parents will complete the Parent-Teacher Relationship Scale II (Vickers & Minke, 1995) to measure the quality of parent-teacher relationships. This 24-item scale includes answer choices from 1 = almost never to 5 = almost always.
Teacher Self-Efficacy for Classroom Behavior Management | Baseline, 4-week, 8-week follow-ups.
  Teachers will complete the Teacher Self-Efficacy Scale - Classroom Management (Tschannen-Moran & Woolfolk Hoy, 2001) measure to rate their self-efficacy in managing classroom behaviors. The 8-item scale ranges from 1 = Nothing to 9= A great deal; higher scores indicate greater self-efficacy.
Teacher Burnout | Baseline, 4-week, 8-week follow-ups.
  Teachers will complete the West Virginia Teacher Burnout Scale (Richmond, Wrench, & Gorham, 2001) to measure teacher burnout. This 20-item scale uses a 5 item Likert scale of 1= strongly disagree to 5= strongly agree. Scores range from 20-80; higher scores indicate greater feelings of burnout.
Racial Awareness, Beliefs, and Attitudes | Baseline, 4-week, 8-week follow-ups.
  Teachers will complete a three-part measure (Fergus, 2016; Neville et al., 2000; Seattle Office of Civil Rights) to assess their racial awareness, beliefs, and attitudes. Part 1 has 10 items and uses a 4-point Likert scale from 1= strongly disagree to 4= strongly agree; part 2 has 20 items and uses a 6-point Likert scale from 1= strongly disagree to 6=strongly agree; part 3 has 12 items and uses a 6-point Likert scale from 1= strongly disagree to 6=strongly agree.
Parent Self-Efficacy | Baseline, 4-week, 8-week follow-ups.
  Parents will complete the Tool to Measure Parenting Self-Efficacy (TOPSE; Kendall & Bloomfield, 2005) subscales of discipline/setting boundaries and control to measure parenting self-efficacy around conflict. The subscales have 6 items each on a 0-10 point scale, and higher scores indicate greater parenting self-efficacy.
Parenting Stress | Baseline, 4-week, 8-week follow-ups.
  Parents will complete the Parental Stress Scale (Berry & Jones, 1995) to measure parental stress. The scale is composed of 18 items, with answers from 1 = strongly disagree to 5 = strongly agree. Scores range from 18-90, with higher scores indicating greater levels of stress.
Top Problems | 4-week and 8-week follow-ups.
  Parents and teachers will complete the Top Problems scale (developed by the investigators) to rate child behavior on the top three behaviors selected to monitor on the Daily Report Card plus overall behavior. Items are scored with a 7-point Likert scale from -3 = much worse to 3 = much better.
Expulsion Risk | Baseline, 4-week, 8-week follow-ups.
  Teachers will complete the Preschool Expulsion Risk Measure (Gilliam and Reyes, 2018) to evaluate perceptions of child expulsion risk. The measure has 12 items, with answer choices on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree.
Implementation Outcomes | 4-week follow-up.
  Participants will complete an Implementation Outcomes survey to evaluate the acceptability, feasibility, and appropriateness of PEAR and provide feedback on potential changes in the procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No